CLINICAL TRIAL: NCT06622213
Title: Comparison of the Efficacy of Mucoadhesive Film with and Without Acmella Oleracea Extract and 0.1% Triamcinolone Acetonide for Treatment of Aphthous Ulcers: a Randomized Control Trial
Brief Title: Mucoadhesive Film With/without Acmella Oleracea & Triamcinolone Acetonide for Aphthous Ulcers
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Kemporn Kitsahawong, Principle investigator, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KKUHE671243; D43DE032294 (NIH)
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Aphthous Stomatitis
Keywords: Oral ulcer
MeSH Terms: conditions — Stomatitis, Aphthous; Oral Ulcer | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: group 1: mucoadhesive film with Acmella oleracea extract, group 2: 0.1% triamcinolone acetonide, and group 3: mucoadhesive film without Acmella oleracea extract.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will not know which treatment each participant will receive (single blinding). Participants will know the type of treatment they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- mucoadhesive film with Acmella oleracea extract (Experimental): Participants received mucoadhesive film with Acmella oleracea extract.
  Interventions: Other: mucoadhesive film with Acmella oleracea extract
- Triamcinolone acetonide (Active Comparator): Participants received 0.1% Triamcinolone acetonide.
  Interventions: Drug: Triamcinolone Acetonide 0.1% Oromucosal Paste
- mucoadhesive film without Acmella oleracea extract (Placebo Comparator): Participants received mucoadhesive film without Acmella oleracea extract.
  Interventions: Other: mucoadhesive film without Acmella oleracea extract

INTERVENTIONS:
Other: mucoadhesive film with Acmella oleracea extract — Apply 1 patch on ulcer 3 times per day (after meals)
  Arms: mucoadhesive film with Acmella oleracea extract
Drug: Triamcinolone Acetonide 0.1% Oromucosal Paste — Apply ¼ inch on ulcer 3 times per day (after meals)
  Other Names: Trinolone oral paste
  Arms: Triamcinolone acetonide
Other: mucoadhesive film without Acmella oleracea extract — Apply 1 patch on ulcer 3 times per day (after meals)
  Arms: mucoadhesive film without Acmella oleracea extract

SUMMARY:
The purpose of this study is to evaluate the effectiveness of mucoadhesive film with or without Acmella oleracea extract compared to standard treatment by using 0.1% triamcinolone acetonide in pain relief, promoting wound healing, healing time and satisfaction in 3 aspects included taste, product used and quality of life after using the product.

DETAILED DESCRIPTION:
Participants who consent and meet the inclusion criteria will be allocated into 3 groups using block randomization: group 1: mucoadhesive film with Acmella oleracea extract, group 2: 0.1% triamcinolone acetonide, and group 3: mucoadhesive film without Acmella oleracea extract.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants aged 18-50 years without any underlying diseases.
2. Participants are voluntary and have signed the informed consent.
3. Participants are literate.
4. Participants can follow the treatment guidelines and follow up.
5. Participants have one untreated oral ulcer lesion.

   * An ulcer has occurred within 48 hours.
   * The ulcer size is less than 10 mm.
   * The ulcer is clearly visible and located on non-keratinized oral mucosa such as buccal mucosa, labial mucosa, alveolar mucosa, or buccal vestibule.
   * The ulcer must be painful.
6. If an ulcer is caused by a denture or orthodontic appliance, the cause must be eliminated before participation.
7. Participants must not be currently participating in any other clinical studies about oral ulcer

Exclusion Criteria:

1. Participants with allergies to herbal extracts, Acmella oleracea, or steroids.
2. Participants with chronic underlying diseases.
3. Participants with underlying diseases that may affect wound healing.
4. Participants receiving anti-analgesic drug, systemic steroids, antibiotics, hormones, NSAIDS, or any drugs that affect the oral mucosa.
5. Oral ulcer lesion larger than 10 mm or lesions resembling herpetic form of aphthous ulcers.
6. Oral ulcers are caused by infection or associated with systemic diseases.
7. Participants with poor oral hygiene requiring emergency treatment.
8. Participants who smoke or consume alcohol regularly.
9. Participants who are pregnant, breastfeeding, or planning to become pregnant during the study period.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Reduction of ulcer size after using product | Base line, day4, day7, day10 and day 14
  Reduction of ulcer size will be evaluated by measuring the diameter of ulcers size using a periodontal probe and photograph on the first day and each follow up visit.
Pain score | Base line, day4, day7, day10 and day 14
  The pain score will be assessed by using a visual analogue scale (VAS) which is a 10-cm line on that was labeled from "no pain"(0) to "worst pain" (10).The pain level will be recorded on the first day. The participants will then reassess their pain score again after receiving the intervention, which will be evaluated at each follow up visit.

SECONDARY OUTCOMES:
Satisfaction score | Day 14
  Participants' satisfaction after using product will be assessed using a visual analogue scale (VAS) which is a 10-cm line on that was labeled from "unsatisfied" (0) to "most satisfied" (10). Satisfaction will be evaluated on the last day of follow-up.
Quality of life score | base line and day 14
  Oral health impact on quality of life will be evaluated using the Thai version of the Oral Health Impact Profile-14 (OHIP-14). The survey classified into 7 dimensions with 2 items per dimension included functional limitation, painful, psychological discomfort, physical disability, psychological disability, social disability, and handicap. Participants must choose the answer based on the frequency of problem occurrence. The frequency level is divided into 5 level: never= 0 point, rarely = 1 point, sometimes = 2 points, often = 3 points, always = 4 points. Total scores in each person range are between 0 to 56 points.The quality of life will be survey on the first and the last day of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Kemporn Kitsahawong, Ph.D, Principal Investigator — KhonKaen university

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ofluoglu D, Ergun S, Warnakulasuriya S, Namdar-Pekiner F, Tanyeri H. An evaluation of the efficacy of a topical gel with Triester Glycerol Oxide (TGO) in the treatment of minor recurrent aphthous stomatitis in a Turkish cohort: A randomized, double-blind, placebo-controlled clinical trial. Med Oral Patol Oral Cir Bucal. 2017 Mar 1;22(2):e159-e166. doi: 10.4317/medoral.21469. PMID 28160585
- [Background] Chatalongkorn, S. (2017). Psychometric Properties of Thai Version of The Oral Health Impact Profile (OHIP-14 Thai). J Prapokklao Hosp Clin Med Educat Center, 34(3), 158-170.